CLINICAL TRIAL: NCT06348901
Title: Clinical Utility of Oxford Cognitive Screen Test to Screen Cognitive Impairment in Post Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Other Study IDs: 2021-09-001; NCT06329232 (obsolete NCT alias)
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects and Stroke patients: Healthy subjects and Stroke patients

SUMMARY:
The goal of this type of study: clinical trial is to assess K-OCS clinical utility in participant population. The main aims:

validate the reliability and validity of the Korean version of the Oxford Cognitive Screen (K-OCS) analyze its sensitivity, specificity, and diagnostic accuracy, and compare its examination participation rates with existing assessment tools to determine the effectiveness of K-OCS in detecting post-stroke cognitive impairment.

ELIGIBILITY:
For stroke patients

1. Inclusion Criteria:

   * Adults over 20 years of age
   * More than 72 hours elapsed since the onset of stroke symptoms.
   * After hearing a detailed explanation of this study and fully understanding it, the subject or legal representative voluntarily decides to participate and agrees in writing to observe the precautions
   * Involved individuals diagnosed with stroke by neurology and rehabilitation medicine specialists based on data acquired from 3T GE Signa System (General Electric, Milwaukee, WI), brain magnetic resonance imaging (MRI), and computed tomography (CT).
2. Exclusion Criteria:

   * Who cannot meet the inclusion criteria

For healthy voluteers

1. Inclusion Criteria:

   * Over 20 years of age
   * A person who is performing an independent daily life
   * A person who voluntarily decides to participate and agrees in writing to abide by the precautions after hearing a detailed explanation of this study and fully understanding it
2. Exclusion Criteria:

   * Who cannot meet the inclusion criteria

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stroke patients and healthy voluteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of K-OCS | Between November 2020 and April 2022
  Measurement of k-ocs is a process of validating K-OCS and assess its clinical utility

SECONDARY OUTCOMES:
Measurement of Korean version of mini-mental state examination (K-MMSE) | Between November 2020 and April 2022
  K-MMSE is a measurement of cognitive level. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe(≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainement and age.
Measurement Korean Version of the Oxford cognitive screen (K-OCS) | Between November 2020 and April 2022
  OCS is an assessment of major cognitive domains of memory, language, number, praxis, executive functions and attention.
Measurement of national institute of health care stroke scale (NIHSS) | Between November 2020 and April 2022
  NIHSS is a measurement for assessing the severity of stroke patients. The scale is made up of 11 different elements that evaluate specific ability. The score for each ability is a number between 0 and 4, 0 being normal functioning and 4 being completely impaired. 42 is the highest score possible, the higher the score, the more impaired a stroke patient is.
Measurement of fuctional independence meausure (FIM) | Between November 2020 and April 2022
  FIM is a measurment to evaluate the funciontional status. FIS is an 18-item including functional capability in six areas of self-care, continence, mobility, transfers, communication and cognition. Each of the 18 items are graded on a scale of 1-7, based on the level of independence in that item

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea